CLINICAL TRIAL: NCT02297087
Title: Next-generation Sequencing of Small Cell Lung Cancer to Identify Actionable Targets for Treatment
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI no longer at site and he does
Sponsor: Western Regional Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: gweiss 13-007
Record Dates: First submitted 2014-11-14; First posted 2014-11-21 (Estimated); Last update posted 2017-11-09 (Actual); Status verified 2017-11

CONDITIONS: Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma

STUDY DESIGN:
Intervention Model Description: This study is testing the specimens for genomic results. There are no other interventions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pilot (Other): Obtain the necessary tumor biopsies to yield sufficient DNA and RNA for Genome-Wide Sequencing (GWS).
  Interventions: Genetic: Standard of care based on target(s) identified via GWS.

INTERVENTIONS:
Genetic: Standard of care based on target(s) identified via GWS.

SUMMARY:
Aim 1 - Launch Pilot Study. In this aim, the investigators seek to launch a pilot study and enroll 12 eligible patients with advanced small cell lung cancer (SCLC) and to obtain the necessary tumor biopsies to yield sufficient DNA and RNA for Genome-Wide Sequencing (GWS).

Aim 2 - Treatment Selection. Completion of this study aim will provide a new clinical paradigm in the treatment of SCLC such that each individual patient would be treated with a single-agent or combination therapy of commercially available agents that relates to particular target(s) that have been identified via GWS.

DETAILED DESCRIPTION:
Participants will be consented into the study after they are found to meet the study inclusion criteria. The clinical staff will schedule a tissue biopsy and a blood draw for the participant. Blood will be sent to Ashion for DNA extraction. Tumor specimens will be shipped to Ashion for DNA and RNA extraction. Ashion will process the samples for DNA and RNA Sequencing in their CLIA certified laboratory. A portion of the nucleic acid will be stored in Ashion and used to confirm actionable targets. Results will be submitted to the physician for possible inclusion in the treatment regimen. After sequencing analysis has been performed, a report will be provided to the treating oncologist. The PI and the treating oncologist may review the results to identify potential treatment. The treating oncologist may use this information at their discretion, and is not required to treat the patient based on the targets identified by the GWS analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients must understand the rigors of the study and provide written informed consent and HIPAA authorization prior to initiation of any study procedures
* Life expectancy > 3 months
* Karnofsky Performance Status ≥ 70
* Diagnosis of histological or cytologically confirmed advanced, incurable SCLC, which has progressed on one or more prior chemotherapeutic, hormonal, or biological regimens for advanced SCLC
* Age ≥ 18 years
* Adequate organ and bone marrow function, defined as: Bone marrow: absolute neutrophil count (ANC) ≥ 1.5 x 109/L; hemoglobin > 9 g/dL; platelets > 100 x 109/L Renal: creatinine clearance ≥ 50 mL/min (calculated according to Cockroft and Gault) or creatinine ≤ 1.5 mg/dL Hepatic: bilirubin ≤ 1.5 x the upper limit of normal (ULN); aspartate transaminases (AST/SGOT) and alanine transaminases (ALT/SGPT) ≤ 2.5 x ULN (or ≤ 5 x ULN if due to underlying liver metastases); internation normalized value for prothrombin time (INR) ≤ 1.5 x ULN (except in the case of anticoagulation therapy), albumin ≥ 2.0
* Good medical candidate for and willing to undergo a biopsy or surgical procedure to obtain tissue, which may or may not be part of the patient's routine care for their malignancy.

Exclusion Criteria:

* Symptomatic CNS metastasis. Patients with a history of CNS metastases, who have been treated, must be stable without symptoms for 4 weeks after completion of treatment, with image documentation required, and must be either off steroids or on a stable dose of steroids for ≥ 2 weeks prior to enrollment
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active serious infection, symptomatic congestive heart failure, unstable angina pectoris, unstable cardiac arrhythmias, psychiatric illness, or situations that would limit compliance with the study requirements or the ability to willingly give written informed consent
* Known HIV, HBV, or HCV infection requiring antiviral therapy.
* Pregnant or breastfeeding patients or any patient of childbearing potential not using adequate contraception.
* Tumor inaccessible for biopsy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
amount of DNA and RNA obtained from tumor biopsies and if can perform Genome-Wide Sequencing (GWS). | 28 Days

CONTACTS AND LOCATIONS:
Overall Officials: Glen Weiss, MD, Principal Investigator — Western Regional Medical Center
Locations (1):
- Cancer Treatment Center of America @ Western Regional Medical Center, Goodyear, Arizona, United States